CLINICAL TRIAL: NCT07311590
Title: A First-in-human Clinical Trial Evaluating the Feasibility of Performing Colonoscopic Polypectomy With a Novel Colonic Intraluminal Endoscopic Support Structure (CIESS) In-situ
Brief Title: A First-in-human Clinical Trial Evaluating a Novel Colonic Intraluminal Endoscopic Support Structure (CIESS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JurongHealth (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2025/1074
Record Dates: First submitted 2025-12-08; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colonoscopy and polypectomy with Colonic Intraluminal Endoscopic Support Structure in-situ (Experimental)
  Interventions: Device: Colonic Intraluminal Endoscopic Support Structure

INTERVENTIONS:
Device: Colonic Intraluminal Endoscopic Support Structure — During colonoscopy, if a left-sided colonic polyps is identified, the colonic intraluminal endoscopic support structure (CIESS) will be deployed. Routine polypectomy will be performed. CIESS will be retrieved after polypectomy is completed. Colonoscopy will be completed as per normal routine.Other Name:

SUMMARY:
The aim of the first-in-human clinical trial is to evaluate the feasibility of performing colonoscopic polypectomy with a novel colonic intraluminal endoscopic support structure (CIESS) in-situ

ELIGIBILITY:
Inclusion Criteria:

* Positive fecal occult blood test

  * ASA I/II
  * only patients with left-sided colonic polyp during colonoscopy will be included into the study eventually

Exclusion Criteria:

* History of malignancy, gastrointestinal tract/ abdominal surgery, diverticular disease, abdominal/ pelvic radiation
* Pregnancy patient
* cognitively impaired patients
* Patients on blood thinners or anticoagulants
* ASA III / ASA IV

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2026-12-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Ability to deploying CIESS in a single attempt | From enrollment to end of treatment at 4 weeks
  Primary outcome measure is whether the CIESS can be deployed successfully in a single attempt - this is a measure of the feasibility of deploying the CIESS during colonoscopy. This outcome will be recorded as "successfully deployed in a single attempt or unsuccessfully deployed in a single attempt"